CLINICAL TRIAL: NCT03814746
Title: A Phase III, Multicenter, Randomized, Double-blind Study to Assess Efficacy and Safety of Two Doses of Crizanlizumab Versus Placebo, With or Without Hydroxyurea/ Hydroxycarbamide Therapy, in Adolescent and Adult Sickle Cell Disease Patients With Vaso-Occlusive Crises (STAND)
Brief Title: Study of Two Doses of Crizanlizumab Versus Placebo in Adolescent and Adult Sickle Cell Disease Patients
Acronym: STAND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSEG101A2301; 2017-001746-10 (EudraCT Number)
Expanded Access: NCT03720626 (Available)
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Sickle Cell Disease; SCD; SEG101; Crizanlizumab; Hydroxyurea/ Hydroxycarbamide Therapy; Vaso-Occlusive Crises; SCA; blood disorders; hemoglobin; red blood cells; sickle-like shape; mutation in hemoglobin gene; sickle-cell trait; sickle-cell crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hematologic Diseases; Sickle Cell Trait | interventions — crizanlizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Crizanlizumab (SEG101) at 5.0 mg/kg (Experimental): Participants received Crizanlizumab (SEG101) at 5.0 mg/kg
  Interventions: Drug: Crizanlizumab (SEG101)
- Crizanlizumab (SEG101) at 7.5 mg/kg (Experimental): Participants received Crizanlizumab (SEG101) at 7.5 mg/kg
  Interventions: Drug: Crizanlizumab (SEG101)
- Placebo (Placebo Comparator): Participants received the placebo drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crizanlizumab (SEG101) — Crizanlizumab was supplied in single use 10 mL glass vials at a concentration of 10 mg/mL. One vial contains 100 mg of crizanlizumab. This is a concentrate for solution for infusion.
  IV.
  Other Names: SEG101
  Arms: Crizanlizumab (SEG101) at 5.0 mg/kg; Crizanlizumab (SEG101) at 7.5 mg/kg
Drug: Placebo — Placebo was supplied in single use 10 mL glass vials at a concentration of 0 mg/mL. This is a concentrate for solution for infusion IV.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 2 doses of crizanlizumab (5.0 mg/kg and 7.5 mg/kg) versus placebo in adolescent and adult sickle cell disease (SCD) patients with history of vaso-occlusive crisis (VOC) leading to healthcare visit.

DETAILED DESCRIPTION:
Study CSEG101A2301 (STAND) is an ongoing Phase III, multicenter, randomized, double-blind study to assess efficacy and safety of two doses of crizanlizumab (5 mg/kg and 7.5 mg/kg) versus placebo, with or without hydroxyurea/ hydroxycarbamide therapy (HU/HC), in adolescent and adult patients with SCD and history of VOC leading to healthcare visit.

This is a multicenter clinical trial comparing 2 doses of crizanlizumab (5 mg/kg and 7.5 mg/kg) versus placebo in addition to standard of care participants might be taking at the time of study start, in adolescent and adult participants with confirmed diagnosis of sickle cell disease (SCD) and history of vaso-occlusive crisis (VOC) leading to a healthcare visit.

240 participants (including 48 adolescents) were planned to be randomized in a 1:1:1 ratio to either 5 mg/kg, 7.5 mg/kg of crizanlizumab or placebo. Randomized participants were stratified by concomitant HU/HC usage (yes/no) and baseline rate of VOCs leading to a healthcare visit in 12 months prior to screening visit (2-4 vs. ≥ 5 VOCs) at the time of enrollment. In November 2020, a capping of 90 adult participants per strata was implemented to ensure adequate opportunity for enrollment into each of the 4 strata.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. Male or female patients aged 12 years and older on the day of signing informed consent. Adolescent include patients aged 12 to 17 years old and adults ≥ 18 years
3. Confirmed diagnosis of SCD by hemoglobin electrophoresis or high performance liquid chromatography (HPLC) [performed locally]. All SCD genotypes are eligible, genotyping is not required for study entry
4. Experienced at least 2 VOCs leading to healthcare visit within the 12 months prior to screening visit as determined by medical history. Prior VOC leading to healthcare visit must resolve at least 7 days prior to Week 1 Day 1 and must include:

   1. Pain crisis defined as an acute onset of pain for which there is no other medically determined explanation other than vaso- occlusion -
   2. which requires a visit to a medical facility and/or healthcare professional,
   3. and receipt of oral/parenteral opioids or parenteral nonsteroidal anti-inflammatory drug (NSAID) analgesia Acute chest syndrome (ACS), priapism and hepatic or splenic sequestration will be considered VOC in this study
5. If receiving HU/HC or L-glutamine (local HA approved medicinal product), must have been receiving the drug for at least 6 months and at a stable dose for at least 3 months prior to Screening visit and plan to continue taking it at the same dose and schedule until the subject has reached one year of study treatment. Patients who have not been receiving such drug must not have received it for at least 6 months prior to Screening visit to be included. Patients must have evidence of insufficient control of acute pain, such as at least one VOC leading to healthcare visit while on HU/HC or L-Glutamine treatment. If receiving erythropoietin stimulating agent, must have been receiving the drug for at least 6 months prior to Screening visit and plan to continue taking the treatment to maintain stable Hb levels at least until the subject has reached one year of study treatment
6. Patients must meet the following central laboratory values prior to Week 1 Day 1:

   * Absolute Neutrophil Count ≥1.0 x 109/L
   * Platelet count ≥75 x 109/L
   * Hemoglobin: for adults (Hb) ≥4.0 g/dL and for adolescents (Hb) ≥5.5 g/dL
   * Glomerular filtration rate ≥ 45 mL/min/1.73 m2 using CKD-EPI formula in adults, and Shwartz formula in adolescents
   * Direct (conjugated) bilirubin < 2.0 x ULN
   * Alanine transaminase (ALT) < 3.0 x ULN
7. ECOG performance status ≤2.0 for adults and Karnofsky ≥ 50% for adolescents

Key Exclusion Criteria:

1. History of stem cell transplant.
2. Participating in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes) and/or planning on undergoing an exchange transfusion during the duration of the study; episodic transfusion in response to worsened anemia or VOC is permitted.
3. Contraindication or hypersensitivity to any drug or metabolites from similar class as study drug or to any excipients of the study drug formulation. History of severe hypersensitivity reaction to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
4. Received active treatment on another investigational trial within 30 days (or 5 half-lives of that agent, whichever is greater) prior to Screening visit or plans to participate in another investigational drug trial.
5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant unless they are using highly effective methods of contraception during dosing and for 15 weeks after stopping treatment.
6. Concurrent severe and/or uncontrolled medical conditions which, in the opinion of the Investigator, could cause unacceptable safety risks or compromise participation in the study.
7. History or current diagnosis of ECG abnormalities indicating significant risk of safety such as:

   * Concomitant clinically significant cardiac arrhythmias (e.g ventricular tachycardia), and clinically significant second or third degree AV block without a pacemaker
   * History of familial long QT syndrome or know family history of Torsades de Pointes
8. Not able to understand and to comply with study instructions and requirements.
9. Received prior treatment with crizanlizumab or other selectin targeting agent

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2026-11-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (5):
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Levine Cancer Insitute Carolinas Healthcare System, Charlotte, North Carolina
  - Univ of Tenn Health Sciences Ctr, Memphis, Tennessee
  - U of TX Health Science Ct, Houston, Texas
- Belgium (3):
  - Novartis Investigative Site, Brussels, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
- Brazil (7):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Valledupar, Cesar Department
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Helsinki, Finland
- France (3):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Accra, Ghana
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- India (2):
  - Novartis Investigative Site, Bhubaneswar, Odisha
  - Novartis Investigative Site, Hyderabad, Telangana
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Irbid, Jordan
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Tripoli
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, The Hague, South Holland
- Novartis Investigative Site, Khoudh, Oman
- Panama (2):
  - Novartis Investigative Site, Panama City, Republica de Panama
  - Novartis Investigative Site, Panama City
- Novartis Investigative Site, Soweto, Gauteng, South Africa
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Adana, Saricam, Turkey (Türkiye)
- United Kingdom (4):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Abboud MR, Cancado RD, De Montalembert M, Smith WR, Rimawi H, Voskaridou E, Guvenc B, Ataga KI, Keefe D, Grosch K, Watson J, Reshetnyak E, Nassin ML, Dei-Adomakoh Y. Crizanlizumab with or without hydroxyurea in patients with sickle cell disease (STAND): primary analyses from a placebo-controlled, randomised, double-blind, phase 3 trial. Lancet Haematol. 2025 Apr;12(4):e248-e257. doi: 10.1016/S2352-3026(24)00384-3. Epub 2025 Mar 12. PMID 40088922
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 240 participants (including 48 adolescents) were planned to be randomized in a 1:1:1 ratio to either 5 mg/kg, 7.5 mg/kg of crizanlizumab or placebo. This study was conducted in 21 countries and 63 centers.
Pre-assignment Details: Screening assessments were done within 1 to 28 days prior to Week 1 Day 1. Re-screening of subjects was only allowed if the subject was not randomized before.
Groups:
- Crizanlizumab (SEG101) at 5.0 mg/kg: Participants received Crizanlizumab (SEG101) 5.0 mg/kg IV infusions on day 1, day 15 and every 4 weeks thereafter.
- Crizanlizumab (SEG101) at 7.5 mg/kg: Participants received Crizanlizumab (SEG101) 7.5 mg/kg IV infusions on day 1, day 15 and every 4 weeks thereafter.
- Placebo: Participants received 0.5mL/kg placebo drug by IV infusions on day 1, day 15 and every 4 weeks thereafter.
Period: Overall Study
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Started | 84 | 83 | 85
Completed (Completed = Ongoing) | 66 | 68 | 58
Not Completed | 18 | 15 | 27
Not completed — Participant decision | 9 | 6 | 15
Not completed — Physician Decision | 2 | 2 | 4
Not completed — Death | 2 | 2 | 2
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 0 | 1 | 2
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 84 | 83 | 85 | 252
Age, Customized [Number; unit: participants]
  Adolescents, 12 - < 18 years | 16 | 18 | 20 | 54
  18 - < 65 years | 68 | 65 | 63 | 196
  65 - < 85 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 49 | 139
  Male | 39 | 38 | 36 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 18 | 60
  Not Hispanic or Latino | 54 | 56 | 57 | 167
  Unknown or Not Reported | 8 | 7 | 10 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 46 | 34 | 43 | 123
  White | 27 | 31 | 26 | 84
  Asian | 6 | 7 | 6 | 19
  American Indian or Alaska Native | 3 | 7 | 6 | 16
  Multiple (White and Black or African American) | 1 | 0 | 0 | 1
  Unknown | 1 | 4 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Vaso-occlusive Crisis (VOC) Events Leading to a Healthcare Visit
Description: VOC is defined as pain crisis (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration.
  Healthcare visit is defined as any visit to a medical facility such as emergency room (ER), hospital and/or office visit, which includes pain management of VOC in situ.
  Annualized rate of corresponding VOC events = (Number of corresponding VOC events * 365)/(number of days in the observation period).
  Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor and erythropoietin therapies to treat SCD and/or to prevent/reduce VOCs), date of randomization + 365 days).
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Mean (Standard Deviation); unit: number of events per year
Groups:
- Placebo: Participants received 0.5mL/kg placebo by IV infusions on day 1, day 15 and every 4 weeks thereafter.
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
number of events per year | 2.5 (2.98) | 1.9 (2.30) | 2.1 (2.81)
Statistical Analysis 1: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; p > 0.999, negative binomial regression model; Rate ratio = 1.08, 95% CI 2-sided [0.76 to 1.55]
Statistical Analysis 2: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; p > 0.999, negative binomial regression model; Rate ratio = 0.89, 95% CI 2-sided [0.62 to 1.27]

2. Secondary Outcome: Annualized Rate of All VOCs Leading to a Healthcare Visit and Treated at Home Over the First-year Post Randomization (Key Secondary)
Description: VOCs are based on documentation by provider following contact with participant. VOC:pain crisis requiring therapy with oral/parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome, priapism and hepatic or splenic sequestration. Healthcare visit:a visit to a medical facility (ER, hospital &/or office visit resulting in pain management of VOC. Managed at home: no visit to any medical facility &/or healthcare professional to receive treatment for VOC. Healthcare contact for medical advice is allowed. Annualized rate of corresponding VOC events = (# of corresponding VOC events * 365)/(# of days in observation period). Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor & erythropoietin therapies to treat SCD &/or to prevent/reduce VOCs), date of randomization + 365 days)
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Mean (Standard Deviation); unit: number of events per year
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
number of events per year | 4.5 (6.49) | 3.1 (2.89) | 3.7 (3.78)
Statistical Analysis 1: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; negative binomial regression model; Rate ratio = 1.21, 95% CI 2-sided [0.87 to 1.70]
Statistical Analysis 2: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; negative binomial regression model; Rate ratio = 0.83, 95% CI 2-sided [0.59 to 1.17]

3. Secondary Outcome: Annualized Rate of All VOCs Leading to a Healthcare Visit and Treated at Home Over 5 Years Post Randomization (Key Secondary)
Description: To compare the efficacy of 5.0 mg/kg vs placebo & 7.5 mg/kg vs placebo on the annualized rate of all VOCs based on documentation by provider following contact with participant. VOC is defined as pain crisis (an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) requiring therapy with oral/parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome, priapism and hepatic or splenic sequestration. Healthcare visit is defined as a visit to a medical facility (emergency room, hospital and/or office visit resulting in pain management of VOC. Managed at home is defined as no visit to any medical facility and/or healthcare professional to receive treatment for VOC. Healthcare contact for medical advice is allowed. The annualized rate of VOC leading to healthcare visit is the number of VOC leading to healthcare visit multiplied by 365 & divided by the number of days in observation period.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Mean Duration of VOCs Leading to a Healthcare Visit Over the First-year Post Randomization
Description: To assess the duration of VOCs leading to healthcare visit in each group. Mean duration of VOC per participant is defined as the average duration of all individual episodes of VOCs leading to healthcare visits of a given participant (a VOC duration is defined as end date of the VOC - start date of the VOC + 1). Participants with no VOC leading to healthcare visits have been excluded.
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization. Participants with no VOC leading to healthcare visits are excluded.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 59 | 52 | 51
days | 7.7 (6.93) | 6.0 (4.54) | 6.6 (5.55)

5. Secondary Outcome: Number of Participants Free From VOCs Leading to a Healthcare Visit Over the First-year Post Randomization
Description: To assess the number of participants free from VOCs leading to healthcare visit.
  VOC is defined as pain crisis (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration. A participant is free from VOC if they do not have a VOC crisis.
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Number; unit: Participants
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
Participants | 25 | 31 | 34

6. Secondary Outcome: Percentage of Participants Free From VOCs Leading to a Healthcare Visit Over the First-year Post Randomization
Description: To assess the percentage of participants free from VOCs leading to healthcare visit. VOC is defined as pain crisis (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration. A participant is free from VOC if they do not have a VOC crisis.
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
Percentage of participants | 29.8 | 37.3 | 40.0

7. Secondary Outcome: Time to First and Second VOCs Leading to a Healthcare Visit Over the First-year Post Randomization
Description: To assess the time to first and second VOC leading to healthcare visit in each group.
  Time to first occurrence of VOC leading to a healthcare visit is defined as the time from the date of randomization to the date of the first occurrence of the VOC.
  Time to second occurrence of VOC leading to a healthcare visit is defined as the time from date of randomization to the date of the second occurrence of VOC.
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization. The estimated time to first and second VOC using Kaplan-Meier analyzed all participants, including those who experienced first (n=59, 52, 51) and second (n=41, 33, 33) events in 5mg/kg, 7.5mg/kg and placebo arms, respectively, those who were at risk, and those who were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
Months
  Time to first occurrence of VOC | 3.9 [2.4 to 6.0] | 6.2 [3.2 to 10.3] | 6.2 [2.8 to 11.9]
  Time to second occurrence of VOC | 10.6 [7.7 to NA] — NA: there were not enough patients or/and events to estimate the upper limit of CI | NA [10.2 to NA] — NA: there were not enough patients or/and events to estimate the median and upper limit of CI | NA [8.9 to NA] — NA: there were not enough patients or/and events to estimate the median and upper limit of CI
Statistical Analysis 1: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; Cox Model; for time to first occurrence of VOC; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.92 to 1.97]
Statistical Analysis 2: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Cox Model; for time to first occurrence of VOC; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.72 to 1.58]
Statistical Analysis 3: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority — for time to second occurrence of VOC; Cox Model; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.81 to 2.04]
Statistical Analysis 4: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Cox Model; for time to second occurrence of VOC; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.59 to 1.54]

8. Secondary Outcome: Annualized Rate of Visits to Clinic, Emergency Room (ER) and Hospitalizations, Both Overall and VOC-related Over the First-year Post-randomization
Description: To assess Healthcare resource utilization (visits to clinic, Emergency room (ER) and hospitalizations) both overall and VOC-related in each group.
  Annualized rate of corresponding healthcare visits =(Number of corresponding healthcare visits * 365)/(number of days in the observation period).
  Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor and erythropoietin therapies to treat SCD and/or to prevent/reduce VOCs), date of randomization + 365 days)
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Mean (Standard Deviation); unit: number of events per year
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
number of events per year
  Annualized rate of all clinic, hospitalizations and ER visits | 3.5 (3.65) | 2.6 (3.21) | 3.0 (3.87)
  Annualized rate of VOC-related clinic, hospitalizations and ER visits | 3.0 (3.52) | 2.2 (3.01) | 2.5 (3.53)
Statistical Analysis 1: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized rate of all visits to clinics, emergency rooms and hospitalizations; Rate ratio = 1.03, 95% CI 2-sided [0.75 to 1.43]
Statistical Analysis 2: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized rate of all visits to clinics, emergency rooms and hospitalizations; Rate ratio = 0.82, 95% CI 2-sided [0.59 to 1.14]
Statistical Analysis 3: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized rate of VOC-related visits to clinics, emergency rooms and hospitalizations; Rate ratio = 1.11, 95% CI 2-sided [0.77 to 1.59]
Statistical Analysis 4: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized rate of VOC-related visits to clinics, emergency rooms and hospitalizations; Rate ratio = 0.87, 95% CI 2-sided [0.60 to 1.25]

9. Secondary Outcome: Annualized Days of Visits to Clinic, Emergency Room (ER) and Hospitalizations, Both Overall and VOC-related Over the First-year Post-randomization
Description: To assess Healthcare resource utilization (visits to clinic, Emergency room (ER) and hospitalizations) both overall and VOC-related in each group.
  Annualized days of corresponding healthcare visits =(Number of days =(Number of days of corresponding healthcare visits * 365)/(number of days in the observation period).
  Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor and erythropoietin therapies to treat SCD and/or to prevent/reduce VOCs), date of randomization + 365 days).
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Mean (Standard Deviation); unit: number of days per year
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
number of days per year
  Annualized days of all clinic, hospitalizations and ER visits | 17.6 (27.80) | 11.3 (14.29) | 12.9 (18.32)
  Annualized days of all VOC-related clinic, hospitalizations and ER visits | 13.8 (18.12) | 9.3 (12.62) | 11.3 (18.35)
Statistical Analysis 1: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized days of all visits to clinics, emergency rooms and hospitalizations; Rate ratio = 1.34, 95% CI 2-sided [0.85 to 2.09]
Statistical Analysis 2: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized days of all visits to clinics, emergency rooms and hospitalizations; Rate ratio = 0.88, 95% CI 2-sided [0.57 to 1.38]
Statistical Analysis 3: Comparison: Crizanlizumab (SEG101) at 5.0 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized days of VOC-related visits to clinics, emergency rooms and hospitalizations; Rate ratio = 1.27, 95% CI 2-sided [0.77 to 2.09]
Statistical Analysis 4: Comparison: Crizanlizumab (SEG101) at 7.5 mg/kg vs Placebo; Test type: Superiority; Negative binomial regression model; for the Annualized days of VOC-related visits to clinics, emergency rooms and hospitalizations; Rate ratio = 0.87, 95% CI 2-sided [0.52 to 1.44]

10. Secondary Outcome: Evolution of Albumin Creatinine Ratio (ACR) Over the First-year Post-randomization (Change From Baseline)
Description: Laboratory values for parameters related to renal function (creatinine, estimated glomerular filtration rate, urine microalbumin, and urine albumin/creatinine ratio) were measured at 6-month intervals over time from baseline.
Time Frame: Over first year post-randomization (Baseline, Week 27 Day 1, Week 51 Day 1)
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Median (Full Range); unit: g/mol
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
g/mol
  Change from baseline at Week 27 Day 1: number analyzed (Participants) | 51 | 64 | 54
  Change from baseline at Week 27 Day 1 | 0.1 [-30 to 96] | -0.0 [-157 to 28] | -0.1 [-20 to 40]
  Chage from baseline at Week 51 Day 1: number analyzed (Participants) | 59 | 58 | 53
  Chage from baseline at Week 51 Day 1 | 0.1 [-34 to 187] | -0.1 [-103 to 49] | -0.2 [-21 to 59]

11. Secondary Outcome: Evolution of Albuminuria (Urine Microalbumin) Over the First-year Post-randomization (Change From Baseline)
Description: as for outcome 10
Time Frame: Over first year post-randomization (Baseline, Week 27 Day 1, Week 51 Day 1)
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Median (Full Range); unit: g/L
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
g/L
  Change from baseline at Week 27 Day 1: number analyzed (Participants) | 65 | 70 | 64
  Change from baseline at Week 27 Day 1 | 0.0 [-1 to 1] | 0.0 [-1 to 0] | 0.0 [-0 to 0]
  Change from baseline at Week 51 Day 1: number analyzed (Participants) | 68 | 64 | 61
  Change from baseline at Week 51 Day 1 | 0.0 [-1 to 1] | 0.0 [-1 to 1] | 0.0 [-0 to 0]

12. Secondary Outcome: Pharmacokinetic (PK) Profile of Crizanlizumab: AUCd15, AUCtau
Description: To characterize the pharmacokinetic (PK) profile of crizanlizumab at 5.0 and 7.5 mg/kg: Area under the (concentration-time profile) curve.
Time Frame: AUCd15 (first-dose) was assessed at W1D1 (pre-dose, 0.5 hr, 2 hrs and 4 hrs post-dose) to W3D1; AUCtau (steady-state) was assessed at W15D1 (pre-dose, 0.5 hr, 2 hrs and 4 hrs post-dose), W15D2, W15D4, W16D1, W17D1, W18D1, W19D1
Population: Pharmacokinetic analysis set 1 includes all participants who provided at least one evaluable PK profile: received the planned treatment at 5 mg/kg or 7.5 mg/kg before single dose PK profile or 3 consecutive doses of the planned treatment before the multiple dose PK profile for the multiple dose PK profile; provided at least one PK parameter; did not have any transfusion of blood product in the last 4 weeks before the first PK sample of the full PK profile, or during the full PK profile.
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg
Number analyzed (Participants) | 76 | 75
hr*ug/mL
  AUCd15 (first dose): number analyzed (Participants) | 64 | 66
  AUCd15 (first dose) | 11300 (2950) | 17000 (4100)
  AUCtau (steady state): number analyzed (Participants) | 44 | 44
  AUCtau (steady state) | 18800 (5470) | 30200 (8580)

13. Secondary Outcome: PK Profile of Crizanlizumab: Cmax
Description: To characterize the pharmacokinetic (PK) profile of crizanlizumab at 5.0 and 7.5 mg/kg: Maximum concentration.
Time Frame: first-dose was assessed at W1D1 (pre-dose, 0.5 hr, 2 hrs and 4 hrs post-dose) through to W3D1; steady-state was assessed at W15D1 (pre-dose, 0.5 hr, 2 hrs and 4 hrs post-dose), W15D2, W15D4, W16D1, W17D1, W18D1, W19D1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg
Number analyzed (Participants) | 76 | 75
ug/mL
  Cmax (first dose): number analyzed (Participants) | 74 | 75
  Cmax (first dose) | 95.9 (29.4) | 143 (45.3)
  Cmax (steady state): number analyzed (Participants) | 47 | 52
  Cmax (steady state) | 108 (60.2) | 162 (57.4)

14. Secondary Outcome: PK Profile of Crizanlizumab: Tmax
Description: To characterize the pharmacokinetic (PK) profile of crizanlizumab at 5.0 and 7.5 mg/kg: Time to maximum concentration.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg
Number analyzed (Participants) | 76 | 75
hr
  Tmax (first dose): number analyzed (Participants) | 74 | 75
  Tmax (first dose) | 2.08 [0.467 to 25.5] | 2.08 [0.500 to 24.2]
  Tmax (steady state): number analyzed (Participants) | 47 | 52
  Tmax (steady state) | 2.00 [0.25 to 24.9] | 3.58 [0.50 to 24.9]

15. Secondary Outcome: PK Profile of Crizanlizumab: Half-life
Description: To characterize the pharmacokinetic (PK) profile of crizanlizumab at 5.0 and 7.5 mg/kg: half life.
Time Frame: steady-state was assessed at W15D1 (pre-dose, 0.5 hr, 2 hrs and 4 hrs post-dose), W15D2, W15D4, W16D1, W17D1, W18D1, W19D1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg
Number analyzed (Participants) | 43 | 43
day | 9.51 (3.67) | 11.2 (3.55)

16. Secondary Outcome: PD Parameter (P-selectin Inhibition)
Description: To characterize the pharmacodynamic (PD) of crizanlizumab at 5.0 and 7.5 mg/kg: P-selectin inhibition (% inhibition multipled by hr)
Time Frame: AUCd15 (first dose): W1D1, W1D2, W1D4, W2D1 and W3D1; steady state: W15D1, W15D2, W15D4, W16D1, W17D1 W18D1 and W19D1
Population: The Pharmacodynamic analysis set 1 includes all participants who provided at least 1 evaluable PD profile: received planned treatment of crizanlizumab at 5 mg/kg or 7.5 mg/kg before single dose PD profile or 3 consecutive doses of planned treatment before the multiple dose PD profile; provided at least 1 PD-AUC (single dose or multiple dose) parameter; did not have any transfusion of blood product in the last 4 weeks before the first PD sample of the full PD profile or during the full PD profile
Measure: Mean (Standard Deviation); unit: h * %
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg
Number analyzed (Participants) | 61 | 63
h * %
  PD-AUCd15 (first dose): number analyzed (Participants) | 55 | 61
  PD-AUCd15 (first dose) | 32700 (3830) | 33100 (3530)
  PD-AUCd29 (steady state): number analyzed (Participants) | 36 | 39
  PD-AUCd29 (steady state) | 65100 (7000) | 66100 (7190)

17. Secondary Outcome: Annualized Rate of Various Subtypes of VOCs Leading to a Healthcare Visit at 1 Year
Description: To compare the efficacy of 5.0 mg/kg versus placebo and 7.5 mg/kg of crizanlizumab versus placebo on the annualized rate of VOCs leading to healthcare visit. VOC is defined as pain crisis which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration. Healthcare visit: any visit to a medical facility such as ER, hospital and/or office visit, which includes pain management of VOC in situ.
  Annualized rate of corresponding VOC events = (Number of corresponding VOC events * 365)/(number of days in the observation period).
  Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor and erythropoietin therapies to treat SCD and/or to prevent/reduce VOCs), date of randomization + 365 days).
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Mean (Standard Deviation); unit: number of events per year
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
number of events per year
  Subtype of VOC: Uncomplicated sickle cell-vaso-occlusive crisis | 2.3 (2.74) | 1.8 (2.27) | 2.0 (2.79)
  Subtype of VOC: Acute chest syndrome | 0.2 (1.44) | 0.0 (0.21) | 0.1 (0.44)
  Subtype of VOC: Hepatic sequestration | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Subtype of VOC: Splenic sequestration | 0.0 (0.00) | 0.0 (0.11) | 0.0 (0.00)
  Subtype of VOC: Priapism | 0.0 (0.00) | 0.0 (0.15) | 0.0 (0.11)

18. Secondary Outcome: Annualized Rate of Various Subtypes of VOCs Leading to a Healthcare Visit at 5 Years
Description: To compare the efficacy of 5.0 mg/kg versus placebo and 7.5 mg/kg of crizanlizumab versus placebo on the annualized rate of VOCs leading to healthcare visit.
  VOC is defined as pain crisis (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration.
  Healthcare visit is defined as any visit to a medical facility such as emergency room, hospital and/or office visit, which includes pain management of VOC in situ.
  The annualized rate of VOC leading to healthcare visit is the number of VOC leading to healthcare visit multiplied by 365 and divided by the number of days in the observation period.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: Annualized Rate of All VOCs Leading to a Healthcare Visit and Treated at Home at 5 Years
Description: To compare the efficacy of 5.0 mg/kg versus placebo and 7.5 mg/kg of crizanlizumab versus placebo on the rates of all VOCs (managed at home + leading to healthcare visit).
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: Number of VOCs Managed at Home at Year 1
Description: To compare the efficacy of 5.0 mg/kg versus placebo and 7.5 mg/kg of crizanlizumab versus placebo on the number of VOC events that were managed at home.
  VOC is defined as pain crisis (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) which requires therapy with oral or parenteral opioids or parenteral NSAID as well as other complicated crisis such as acute chest syndrome (ACS), priapism and hepatic or splenic sequestration. Managed at home is defined as no visit to any medical facility and/or healthcare professional to receive treatment for VOC. Healthcare contact for medical advice was allowed.
Time Frame: 1 year
Population: The FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Number; unit: total number of VOC events
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg | Crizanlizumab (SEG101) at 7.5 mg/kg | Placebo
Number analyzed (Participants) | 84 | 83 | 85
total number of VOC events | 163 | 106 | 129

21. Secondary Outcome: Number of VOCs Managed at Home at 5 Years
Description: as for outcome 20
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

22. Secondary Outcome: Absolute Change From Baseline in Hemoglobin
Description: To assess safety of crizanlizumab over the study period.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

23. Secondary Outcome: Growth and Sexual Maturity Assessment in Adolescents (Tanner Stage)
Description: To assess safety of crizanlizumab over the study period.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

24. Secondary Outcome: Immunogenicity: Measurement of Anti-drug Antibodies (ADA) to Crizanlizumab
Description: To assess immunogenicity of crizanlizumab over the study period.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: This primary analysis report includes data with a cut-off date 31-Aug-2022. Adverse events and deaths were collected from first dose of study treatment to105 days post-last infusion (defined as on-treatment), up to max on-treatment period of approx. 5 years.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Groups:
- Crizanlizumab (SEG101) at 5.0 mg/kg (On-treatment); Crizanlizumab (SEG101) at 7.5 mg/kg (On-treatment); Placebo (On-treatment): AEs during on-treatment period (up to 105 days post-last infusion)
Arm/Group | Crizanlizumab (SEG101) at 5.0 mg/kg (On-treatment) | Crizanlizumab (SEG101) at 7.5 mg/kg (On-treatment) | Placebo (On-treatment)
All-Cause Mortality (participants affected / at risk) | 2/84 | 2/83 | 2/85
Serious Adverse Events (participants affected / at risk) | 35/84 | 22/83 | 26/85
Other Adverse Events (participants affected / at risk) | 67/84 | 71/83 | 66/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab (SEG101) at 5.0 mg/kg (On-treatment) (N=84) | Crizanlizumab (SEG101) at 7.5 mg/kg (On-treatment) (N=83) | Placebo (On-treatment) (N=85)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Bone marrow necrosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 2 | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 1 | 1
Epiretinal membrane (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Ulcer (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 5 | 6 | 4
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 5 | 1
Sepsis (Infections and infestations) | 3 | 1 | 2
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab (SEG101) at 5.0 mg/kg (On-treatment) (N=84) | Crizanlizumab (SEG101) at 7.5 mg/kg (On-treatment) (N=83) | Placebo (On-treatment) (N=85)
Anaemia (Blood and lymphatic system disorders) | 3 | 8 | 4
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 5 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 8
Constipation (Gastrointestinal disorders) | 8 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 7
Nausea (Gastrointestinal disorders) | 14 | 8 | 8
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 5
Vomiting (Gastrointestinal disorders) | 7 | 8 | 4
Chest pain (General disorders) | 5 | 7 | 7
Fatigue (General disorders) | 6 | 11 | 3
Pyrexia (General disorders) | 22 | 17 | 22
COVID-19 (Infections and infestations) | 16 | 21 | 14
Gastroenteritis (Infections and infestations) | 3 | 6 | 4
Influenza (Infections and infestations) | 5 | 3 | 3
Nasopharyngitis (Infections and infestations) | 4 | 5 | 6
Pneumonia (Infections and infestations) | 6 | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 0
Urinary tract infection (Infections and infestations) | 9 | 8 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 2 | 3
Alanine aminotransferase increased (Investigations) | 6 | 2 | 1
SARS-CoV-2 test positive (Investigations) | 4 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 17 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 16
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 10 | 13
Dizziness (Nervous system disorders) | 6 | 2 | 2
Headache (Nervous system disorders) | 21 | 13 | 15
Insomnia (Psychiatric disorders) | 4 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03814746/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03814746/SAP_001.pdf